CLINICAL TRIAL: NCT01188954
Title: Randomized Clinical Trial of Doxycycline Versus Standard Care to Prevent Seroma Formation at Femoral Artery/Vein Cannulation Site After Cardiopulmonary By-Pass
Brief Title: Doxycycline Versus Standard Care to Prevent Seroma Formation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment process was slower than expected.
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, John P Nabagiez, MD, M.D., Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Doxy 10-006
Record Dates: First submitted 2010-06-22; First posted 2010-08-26 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Seroma
Keywords: Seroma; Doxycycline; Cardiopulmonary By-Pass; Femoral Artery/Vein Cannulation; Prevent Seroma Formation
MeSH Terms: conditions — Seroma | interventions — Doxycycline; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxycycline (Active Comparator): Doxycyline, family of tetracycline antibiotics, used to scleroses the lymphatic vessels that may have transected during dissection.
  Interventions: Drug: doxycycline
- Normal Saline/Water (Placebo Comparator): The standard care is wetting and suctioning fluids followed with suturing of the groin.
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: doxycycline — 50 ml/mg
  Arms: Doxycycline
Other: No intervention — Normal Saline/Water
  Other Names: Normal Saline, Sterile Water
  Arms: Normal Saline/Water

SUMMARY:
A seroma is a collection of fluid other than pus or blood which forms through the division of numerous lymphatic channels, which normally drain the interstitial space under the skin. These channels become disrupted during surgical procedure and lead to seroma formation. This collection of fluid causes pressure in the local area, patient discomfort, and provides unfortunately an excellent culture medium for bacteria. Seroma development has been previously described in femoral vessel groin cannulation dissections after surgery. Conventional therapy is limited to draining the fluid, sometimes more than once, until there is full resolution of the seroma. If fluid collection recurs at the surgical site, sclerosant therapy with agents such as doxycycline. Doxycycline has been found to be a cost effective agent used as a sclerosant, which belongs to tetracycline class of antibiotics. The investigators hypothesize that prophylactic use of doxycycline at the site of femoral cannulation will prevent or minimize the area of seroma formation as compared to standard care of patients. The aim is driven towards limiting patient discomfort and visits to the clinic and to improve clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Male and female candidates (>18 and <85 years of age) undergoing Cardiopulmonary By-Pass via Femoral/Groin access as part of their routine cardiothoracic scheduled procedure will be approached for their interest in participation in the study.

Exclusion Criteria:

* A history of allergic reaction to doxycycline (Adoxa, Doryx, Oracea, Vibramycin) or any classes of tetracyclines- demeclocycline (Declomycin), or minocycline (Dynacin, Minocin, Solodyn, Vectrin).
* Patients who are not undergoing Cardiopulmonary By-Pass through femoral access.
* Active infection in the groin region.
* Females who are pregnant or lactating and breast feeding.
* Who do not wish to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
evaluate the efficacy of doxycycline in the prevention of the complication of seroma post-cannulation | 1 year
  The primary aim of this study is to evaluate the efficacy of doxycycline in the prevention of the complication of seroma post-cannulation for cardiopulmonary bypass via femoral access, when compared to standard care.

SECONDARY OUTCOMES:
Identification of predictors of response and complication | 1 year
  The secondary aims include identification of predictors of response and complication, and success rates, as well as, assessment of clinical outcome and Health-Well Being

CONTACTS AND LOCATIONS:
Overall Officials: Kourosh T Asgarian, DO, Principal Investigator — Staten Island University Hospital
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States

REFERENCES:
- [Background] Caliendo MV, Lee DE, Queiroz R, Waldman DL. Sclerotherapy with use of doxycycline after percutaneous drainage of postoperative lymphoceles. J Vasc Interv Radiol. 2001 Jan;12(1):73-7. doi: 10.1016/s1051-0443(07)61407-9. PMID 11200357
- [Background] Swan MC, Furniss D, Cassell OC. Surgical management of metastatic inguinal lymphadenopathy. BMJ. 2004 Nov 27;329(7477):1272-6. doi: 10.1136/bmj.329.7477.1272. No abstract available. PMID 15564260
- [Background] Heffner JE, Standerfer RJ, Torstveit J, Unruh L. Clinical efficacy of doxycycline for pleurodesis. Chest. 1994 Jun;105(6):1743-7. doi: 10.1378/chest.105.6.1743. PMID 8205870